CLINICAL TRIAL: NCT03383146
Title: A 52-week, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Evaluate the Safety and Efficacy of Relamorelin in Patients With Diabetic Gastroparesis
Brief Title: A Safety and Efficacy Study of Relamorelin in Diabetic Gastroparesis Study 04
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Relamorelin program is being terminated solely based on a business decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RLM-MD-04; 2017-002144-33 (EudraCT Number)
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Gastroparesis; Diabetes Mellitus
Keywords: diabetic gastroparesis; vomiting
MeSH Terms: conditions — Gastroparesis; Diabetes Mellitus; Vomiting | interventions — relamorelin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo injected subcutaneously twice daily for up to 52 weeks. De novo (New) participants, who did not participate in the previous relamorelin studies, began the study with a 2-week placebo run-in.
  Interventions: Drug: Placebo
- Relamorelin 10 μg (Experimental): Relamorelin 10 micrograms (μg) injected subcutaneously twice daily for up to 52 weeks. De novo (New) participants, who did not participate in the previous relamorelin studies, began the study with a 2-week placebo run-in.
  Interventions: Drug: Relamorelin

INTERVENTIONS:
Drug: Placebo — Placebo injected subcutaneously twice daily.
  Arms: Placebo
Drug: Relamorelin — Relamorelin 10 μg injected subcutaneously twice daily.
  Arms: Relamorelin 10 μg

SUMMARY:
A 52-week study to compare the efficacy of relamorelin with that of placebo in participants with diabetic gastroparesis (DG) with respect to the core signs and symptoms of diabetic gastroparesis.

ELIGIBILITY:
Inclusion Criteria:

Two different groups of participants may enter into the study:

1. Rollover Participants

   Participants who were not randomization-eligible at the end of the Run-in Period of lead-in studies RLM-MD-01 (NCT03285308) or RLM-MD-02 (NCT03426345) are eligible to be randomized in the study if all of the following criteria apply:

   •In the lead-in studies, participants must have met all screening visit and Run-in Period criteria for randomization into the Treatment Period (including compliance with dosing, entry of diary data into the Diabetic Gastroparesis Symptom Severity Diary (DGSSD)) except that:
   * They had zero vomiting episodes and an average daily Diabetic Gastroparesis Symptom Severity Score (DGSSS) of ≥12 at the end of the lead-in study Run-in Period, as reported using the electronic hand-held device; OR
   * They had vomiting episodes and an average daily DGSSS of ≥12 but <16 at the end of the lead-in study Run-in Period, as reported using the electronic hand-held device
2. De Novo Participants

   * Type 1 Diabetes Mellitus (T1DM) or Type 2 Diabetes Mellitus (T2DM) of at least 5 years' duration, with controlled and stable blood glucose levels and hemoglobin A1c (HBA1c) ≤11%
   * DG defined as at least a 3-month history prior to Screening of symptoms (one of which must be nausea) on an ongoing basis that are suggestive of gastroparesis (GP) (e.g., nausea, abdominal pain, postprandial fullness, bloating, vomiting, and early satiety)
   * Compliance with the entry of data into the hand-held electronic device during the Run-in Period
   * Compliance with administration of subcutaneous (SC) twice daily injections during the Run-in Period
   * The average of the daily DGSSS from the 2-week, Run-in Period must be ≥12

Exclusion Criteria:

1. Both Rollover and De Novo Participants

   •Participants with a known allergy or hypersensitivity to the study treatments and their excipients (i.e., mannitol or phenol)
2. Rollover Participants

   •Participants will be excluded from this study if any of the lead-in study exclusion criteria apply at the Screening Visit and at the end of the Run-in Period for randomization into the Treatment Period of studies RLM-MD-01 and RLM-MD-02, except as specified in the inclusion criteria
3. De Novo Participants

   * History of anorexia nervosa, binge-eating, bulimia, or other eating disorder within 5 years of the Screening Visit
   * History of intestinal malabsorption or pancreatic exocrine insufficiency
   * History of belching disorders, other nausea and vomiting disorders
   * Gastric or duodenal ulcer within 3 months of Screening
   * History of malignancy in the 3 years prior to Screening, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
   * Currently receiving parenteral feeding or presence of a nasogastric or other enteral tube for feeding or decompression
   * Use of metoclopramide, domperidone, prucalopride, macrolide antibiotics (e.g., erythromycin, clarithromycin, azithromycin), or other drugs considered to be GI promotility agents for at least 10 days prior to the start of the Run-in Period
   * Currently taking opiates, or expecting to use opiates during the course of the clinical study
   * Treatment with glucagon-like peptide-1 (GLP-1) agonist for at least 6 weeks prior to the start of the Run-in Period
   * History of pyloric injection of botulinum toxin within 6 months of screening
   * History of gastric surgery such as fundoplication, gastrectomy, gastric pacemaker placement, vagotomy, or bariatric procedure (a history of diagnostic endoscopy is not exclusionary)
   * Randomization in any previous study in which relamorelin was a treatment
   * Allergic to, or intolerant of egg, wheat, milk, or algae, as these are components of the gastric emptying breath test (GEBT) study meal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvy Schneier, Study Director — Allergan
Locations (348):
- United States (182):
  - Pinnacle Research Group, Anniston, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - Simon Williamson Clinic, Birmingham, Alabama
  - Digestive Health Specialist of the South East, Dothan, Alabama
  - G & L Research, LLC, Foley, Alabama
  - Avant Research Associates, Huntsville, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Phoenix Clinical LLC., Phoenix, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Synexus Clinical Research US, Inc., Tucson, Arizona
  - Preferred Research Partners, Inc., Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - Unity Health - Searcy Medical Center, Searcy, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - GW Research Inc, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Aurora Care Clinic, LLC, Costa Mesa, California
  - TriWest Research Associates, El Cajon, California
  - Diagnamics Inc., Encinitas, California
  - VVCRD Research, Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Angel City Research Inc., Los Angeles, California
  - Stanford Hospital, Palo Alto, California
  - Optimal Research California, San Diego, California
  - Medical Associates Research Group, Inc, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Upland Clinical Research, Upland, California
  - Synexus Clinical Research US, Inc., Vista, California
  - New Hope Research Development, Whittier, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Synexus, Colorado Springs, Colorado
  - Gastroenterology Associates of Fairfield County, P.C., Bridgeport, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Innovative Research of West FL, Inc., Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - ALL Medical Research, LLC, Cooper City, Florida
  - Top Medical Research, Cutler Bay, Florida
  - Palmetto Research, LLC, Hialeah, Florida
  - Vida Clinical Trials, Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - APF Research LLC, Miami, Florida
  - AMPM Research Clinic, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - American Research Institute, Inc, Miami, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Synexus, Pinellas Park, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Gwinnett Research Institute, LLC, Buford, Georgia
  - Summit Clinical Research, LLC., Carnesville, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - Clinical Research Consultants of Atlanta, Suwanee, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - North Shore University Health System, Evanston, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Synexus Clinical Research US, Inc., Evansville, Indiana
  - American Research, LLC, Jeffersonville, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Health Science Research Center, Pratt, Kansas
  - WestGlen Gastrointestinal Consultants, Shawnee Mission, Kansas
  - Cotton-O'Neil Clinical Research Center - Digestive Health, Topeka, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Via Christi Clinic, PA, Wichita, Kansas
  - St. Elizabeth Healthcare â€" Clinical Research Institute, Erlanger, Kentucky
  - University of Louisville, Louisville, Kentucky
  - WK Physicians Network, Bossier City, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - Cronola LLC, Houma, Louisiana
  - Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Clinical Trials of America, Inc., West Monroe, Louisiana
  - Metropolitan Gastroenterology Group PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Frederick Gastroenterology Associates, PA an Elligo Health Research Site, Frederick, Maryland
  - Woodholme Gastroenterology Associates, P.A., Glen Burnie, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Vida Clinical Studies, Dearborn, Michigan
  - Aa Mrc, Llc, Flint, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Gastroenterology Associates of Western Michigan, West Michigan Clinical Research Center, Wyoming, Michigan
  - MNGI Digestive Health, Coon Rapids, Minnesota
  - Synexus Clinical Research US, Inc., Richfield, Minnesota
  - Synexus Clinical Research US, Inc, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - Diabetes and Endocrine Associates, P.C., Omaha, Nebraska
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Clinical Research of South Nevada - CROSN, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Garden State Endocrinology LLC, Brick, New Jersey
  - Synexus Clinical Research US, Inc., Bridgeton, New Jersey
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - United Health Services Hospitals, Inc., Johnson City, New York
  - CHEAR Center LLC, The Bronx, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Carolinas Healthcare-Charlotte, Charlotte, North Carolina
  - Carolina Digestive Health Associates, PA, Concord, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Vidant Multispeciality Clinic - Kinston, Kinston, North Carolina
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - PMG Research Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - Dayton Gastroenterology,Inc., Beavercreek, Ohio
  - Diabetes & Endocrinology Associates of Stark County, Inc., Canton, Ohio
  - Synexus Clinical Research US - Cincinnati, Cincinnati, Ohio
  - Synexus Clinical Research US, Inc, Cincinnati, Ohio
  - Endocrinology Research Associates, Inc., Columbus, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - CIC America Clinical Inquest Center Ltd., Dayton, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Premier Clinical Research d.b.a. STAT Research, Franklin, Ohio
  - Family Practice Center of Wadsworth, Inc., Wadsworth, Ohio
  - Centennial Health-Synexus, Oklahoma City, Oklahoma
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Family Medical Associates, Research Department, Levittown, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Synexus Clinical Research US, Inc, Anderson, South Carolina
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Carolina Medical Research, Clinton, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Synexus Clinical Research, Greer, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinsearch, Chattanooga, Tennessee
  - Gastroenterology Centers of the Midsouth, Germantown, Tennessee
  - East Tennessee Research Institute, Johnson City, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - DiscoveResearch, Inc., Beaumont, Texas
  - ClinRx Research, LLC, Carrollton, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Biopharma Informatic Inc., Research Center, Houston, Texas
  - Houston Endoscopy and Research Center, Inc., Houston, Texas
  - Rodriguez Clinical Trials, Houston, Texas
  - Amir Hassan, MD, PA, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Sagact Pllc., San Antonio, Texas
  - Synexus Clinical Research US, Inc., San Antonio, Texas
  - Synexus Clinical Research US, Inc., Layton, Utah
  - Synexus Clinical Research US, Inc., Murray, Utah
  - Advanced Research Institute, Inc., Ogden, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Verity Research Inc., Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Manassas Clinical Research Centre, Manassas, Virginia
  - VA Medical Center McGuire VAMC, Richmond, Virginia
  - Washington Gastroenterology PLLC, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Argentina (10):
  - Consultorios Asociados de Endocrinologia e InvestigaciÃ³n Cl, Buenos Aires, Buenos Aires
  - Hospital Sirio Libanes, CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata SRL, Mar del Plata, Buenos Aires
  - CIPREC, Buenos Aires, Ciudad Autonoma deBuenos Aires
  - Instituto de Investigaciones Clinicas de Rosario, Rosario, Santa Fe Province
  - Instituto Medico Catamarca-I.ME.C, Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Centro Universitario de Investigacion en Farmacologia Clinic, Corrientes
  - Instituto Privado de Investigaciones Clinicas de Cordoba, Córdoba
  - CIDIM - Centro Integral de Diagnóstico por Imágenes Marchegian, Córdoba
- Australia (3):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital - Central Adelaide Local Health Network Incorporated, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (4):
  - Ordination, Osterreicher, Styria
  - VIVIT Institute, am LKH Feldkirch, Feldkirch, Vorarlberg
  - Privatklinik wehlre-Diakonissen, Salzburg
  - Oö. Gesundheits- und Spitals-AG/LKH Steyr, Steyr
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen, Gastro-Enterologie,, Edegem, Antwerp
  - UZ Brussel, Jette, Brussels Capital
  - AZ Sint Lucas Brugge, Bruges, West-Vlaanderen
- Brazil (10):
  - Hospital Universitário Walter Cantídio, Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Hospital Universitário João de Barros Barreto - UFPA, Belém, Pará
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Instituto Catarinense de Endocrinologia e Diabetes (ICED), Joinville, Santa Catarina
  - Scentryphar Pesquisa Clínica Ltda, Campinas, São Paulo
  - Instituto de Pesquisa Clinica em Campinas, Campinas, São Paulo
  - Instituto de Estudos e Pesquisas Clinicas do Ceara IEP/CE - Oncology, Fortaleza
  - IPEC-Instituto de Pesquisa Clinica, São Paulo
  - CPQuali Pesquisa Clinica Ltda, São Paulo
- Bulgaria (4):
  - MHAT Yuliya Vrevska Byala, Byala, Ruse
  - UMHAT - Kaspela- EOOD, Plovdiv
  - Medical Center Asklepion - Humane Medicine Research EOOD, Sofia
  - Alexandrovska University Hospital, Sofia
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - Central Alberta Research Centre, Red Deer, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Patient research centre, St. John's, Newfoundland and Labrador
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
  - Recherche GCP Research, Montreal, Quebec
- Colombia (11):
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Centro Cardiovascular Colombiano Clínica Santa María, Medellín, Antioquia
  - Centro Cardiovascular y de Diabetes, Barranquilla, Atlántico
  - Fundación del Caribe para la InvestigacionBiomédica-Fundación BIOS, Barranquilla, Atlántico
  - Medplus Centro de Recuperacion Integral S.A.S., Bogotá, Bogota D.C.
  - Endocare Ltda., Bogotá, Bogota D.C.
  - Asociación Colombiana de Diabetes, Bogotá, Cundinamarca
  - Healthy Medical Center, Zipaquirá, Cundinamarca
  - Centro de Investigaciones Clínicas IPS CARDIOMET Pereira, Pereira, Risaralda Department
  - IPS Centro Medico Julian Coronel S.A, Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A., Cali, Valle del Cauca Department
- Denmark (2):
  - Steno Diabetes Center Copenhagen, Hellerup, Copenhagen
  - Gastroenheden, Hvidovre hospital, Hvidovre, København
- Germany (6):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-Wurttemberg
  - Studienzentrum Schwittay, Böhlen, Saxony
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Clinical Research Hamburg, Hamburg
  - Israelitisches Krankenhaus, Hamburg
  - KRH Klinikum Siloah, Hanover
- Hungary (5):
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger, Heves County
  - Hetenyi Geza Hospital, Szolnok, Jász-Nagykun-Szolnok
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg, Zala County
  - Strázsahegy Gyógyszertár Medicina, Budapest
  - Szegedi TudomanyegyetemSzent-Gyorgyi Albert Klinikai Kozpont és Altalanos Orvostudomanyi Kar Belgyogyaszati Klinika, Szeged
- India (22):
  - Kumudini Devi Diabetes Research Center; Ramdevrao Hospital, Hyderabad, Andhra Pradesh
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Dr. Jivraj Mehta Smarak Health Foundation Bakeri Medical Research Centre - Gasterentrology, Ahmedabad, Gujarat
  - Zydus Hospital, Ahmedabad, Gujarat
  - Lifecare Clinic and Research Centre - Internal Med/Diabetology, Bangalore, Karnataka
  - Diacon Hospital and research Center - Diabetology, Bengaluru, Karnataka
  - Victoria Hospital Bangalore Medical College and Research Institute, Bengaluru, Karnataka
  - Rajalakshmi Hospital, Bengaluru, Karnataka
  - Bhatia Hospital, Mumbai, Maharashtra
  - B. J. Government Medical College and Sassoon General Hospitals, Pune, Maharashtra
  - Universal Hospital, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - S R Kalla (SRK) Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Marudhar Hospital, Jaipur, Rajasthan
  - Eternal Hospital - Diabetology, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - M.V. Hospital for Diabetes & Diabetes Research Centre, Chennai, Tamil Nadu
  - Kovai Diabetes Speciality Centre, Coimbatore, Tamil Nadu
  - Arthur Asirvatham Hospital, Madurai, Tamil Nadu
  - M V Hospital & Research Centre, Lucknow, Uttar Pradesh
  - Sir Ganga Ram Hospital (SGRH), Delhi
  - Vinaya Hospital & Research Centre, Mangalore
- Bnei-Zion MC, Haifa, Israel
- Latvia (4):
  - Kraslava Hospital, Krāslava, Kraslavas Nov.
  - Polana-D, Daugavpils
  - Pauls Stradins Clinical University Hospital, Endokrinologijas nodala, Riga
  - Digestive Diseases Centre GASTRO, Riga
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - Clinical Investigation Centre, Kuala Lumpur
  - Clinical Trial Unit, School of Medical Sciences, Health Campus, Hospital Universiti Sains Malaysia, Kubang Kerian
  - Hospital Taiping, Taiping
- Mexico (13):
  - Unidad de Investigacion Clinica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Consultorio particular, Guadalajara, Jalisco
  - Unidad de Investigación Clínica en Medicina S.C/, Guadalajara, Jalisco
  - Clinicos Asociados BOCM SC, Mexico City, Mexico City
  - Mentrials Sa de Cv, Mexico City, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Prevencion de E - Endocrinology, Mexico City, Mexico City
  - Centro de Atención e Investigación en Factores de Riesgo Car, Mexico City, Mexico City
  - Centro de Desarrollo Biomédico S.C.P, Mérida, Yucatán
  - Centro de Investigacion Cardiometabolica de Aguascalientes SA de CV, Aguascalientes
  - Hospital Cardiologica Aguascalientes, Aguascalientes
  - Dioderm Instituto de Investigacion, Durango
  - CIADEN (Centro de Investigación y Atención de Diabetes, Endocrinología y Nutrición), Durango
  - Sociedad de Metabolismo y Corazon S.C., Veracruz
- Philippines (7):
  - West Visayas State University Medical Center, Iloilo City, IloIlo
  - Manila Doctors Hospital, Ermita, Manila, Metropolitan Manila
  - San Juan De Dios Educational Foundation, Inc., Pasay, Metropolitan Manila
  - Cardinal Santos Medical Center, San Juan City, National Capital Region
  - Ospital ng Makati, Makati City, NCR
  - Perpetual Succor Hospital, Cebu City
  - St. Luke's Medical Center, Quezon City
- Poland (3):
  - Specjalistyczny Gabinet Neurologiczny Marta Banach, Krakow, Lesser Poland Voivodeship
  - CenterMed Krakow Ltd, Krakow, Malopolska
  - Centrum Medyczne Lukamed, Chojnice
- Russia (4):
  - Saint-Petersburg City Pokrovskaya Hospital, St-Petersburg, Leningradskaya Oblast'
  - GUZ Saratov City Clinical Hospital 9, Saratov, Saratov Oblast
  - Scientific Institute of Clinical and Experimental Lymphology, Novosibirsk
  - Rostov on Don, Rostov-on-Don
- Singapore (3):
  - National University Hospital, Singapore
  - Changi General Hospital, Singapore
  - Singapore General Hospital, Singapore
- South Africa (5):
  - FARMOVS, Bloemfontein, Free State
  - Wits Clinical Research, Johannesburg, Gauteng
  - Synexus Stanza Clinical Research Centre, Pretoria, Gauteng
  - Watermeyer Clinical Research Site, Pretoria, Val de Grace
  - Synexus Helderberg Clinical Research Centre, Somerset West
- South Korea (3):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Sanggye Paik Hospital, Inje University College of Medicine, Seoul, Nowon-gu
  - Asan Medical Center, Seoul
- Hospital Universitario Principe de Asturias, Madrid, Spain
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Ukraine (16):
  - State Institution Ukrainian State Research Institute of Medical and Social Problems of Disability of the Ministry of Health of Ukraine, Dnipro, Dnipropetrovsk Oblast
  - Municipal Institution, City Hospital #7, polyclinic department, c. Zaporizhzhia, Zaporizhzhia, Zaporizhzhia Oblast
  - Chernivtsi Regional Clinical Hospital, Chernivtsi
  - Regional Municipal noncommercial Enterprise "Chernivtsi Regional Endocrinology Center", Polyclinic department, Higher State Educational Establishment of Ukraine "Bukovinian State Medical University", Department of Clinical Immunology, Allergology and Endo, Chernivtsi
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Municipal nonprofit entity of Kharkiv municipal council, Kharkiv
  - Clinical Endocrinology of SI "V.Danilevsky Institute for endocrine pathology problems National Academy of Medical sciences of Ukraine", Kharkiv
  - Communal Institution Kherson City Clinical Hospital, Kherson
  - Kyiv Railway Clinical Hospital No-2 of Branch of Healthcare Center of the PJSC Ukrainian Railway , Endocrynology Department, Kyiv
  - Polyclinic of medical services and rehabilitation department of State Joint-Stock Holding Company Artem, day-patient unit, Kyiv
  - Odessa Railway Clinical Hospital of Branch of HC JSC Ukrzaliznytsia, Odessa National Medical University, Odesa
  - Poltava Regional Clinical Hospital, Poltava
  - Private Small-Scale Enterprise Medical Centre Pulse, Vinnytsia
  - Vinnytsia Regional Clinical highly specialized Endocrinology Centre, Vinnytsia
  - Municipal Institution 6th City Clinical Hospital, Dept of Gastroenterology, Zaporizhzhia
- United Kingdom (11):
  - Biomedical Research Centre, Nottingham, East Midland
  - MAC Clinical Research Manchester, Manchester, Greater Manchester
  - Royal Oldham Hospital, Oldham, Lancashire
  - MAC Clinical Research, Liverpool, Merseyside
  - MAC Research, Exchange House, Cannock, Staffordshire
  - University Hospitals of North Midlands, Stoke-on-Trent, Staffordshire
  - MAC Clinical Research, Monarch House, Leeds, West Yorkshire
  - MAC Research, Barnsley
  - MAC Clinical Research, Kaman Court, Blackpool
  - Mid Essex Hospital Services NHS Trust Broomfield Hospital, Chelmsford
  - MAC Clinical Research, GAC House, Manchester

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the placebo run-in of relamorelin studies: RLM-MD-01 [NCT03285308] and RLM-MD-02 [NCT03426345] were eligible to rollover to this study. De novo (New) participants, who had not participated in the previous studies, were also eligible for enrollment.
Period: Overall Study
Arm/Group | Placebo | Relamorelin 10 μg
Started | 148 | 302
Safety Population (Safety Population included all participants who received ≥1 administration of study treatment.) | 145 | 299
Run-in Period (Run-in Period included rollover participants from previous relamorelin study RLM-MD-01 or RLM-MD-02 who met all the inclusion and exclusion criteria.) | 91 | 207
Completed | 63 | 118
Not Completed | 85 | 184
Not completed — Screen Failure | 1 | 0
Not completed — Adverse Event | 6 | 18
Not completed — Lack of Efficacy | 0 | 3
Not completed — Withdrawal by Subject | 20 | 36
Not completed — Lost to Follow-up | 5 | 15
Not completed — Death | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Deviation | 1 | 8
Not completed — Study Terminated by the Sponsor | 48 | 95
Not completed — Reason not Specified | 4 | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all randomized participants.
Groups:
- Relamorelin 10 μg: Relamorelin 10 μg injected subcutaneously twice daily for up to 52 weeks. De novo (New) participants, who did not participate in the previous relamorelin studies, began the study with a 2-week placebo run-in.
- Total: Total of all reporting groups
Arm/Group | Placebo | Relamorelin 10 μg | Total
Number analyzed (Participants) | 148 | 302 | 450
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (12.37) | 57.9 (11.57) | 57.6 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 224 | 326
  Male | 46 | 78 | 124
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 82 | 132
  Not Hispanic or Latino | 98 | 220 | 318
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 11 | 18
  Asian | 0 | 9 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 27 | 53 | 80
  White | 109 | 218 | 327
  More than one race | 4 | 11 | 15
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Diabetic Gastroparesis Symptom Severity Score (DGSSS)
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the Diabetic Gastroparesis Symptom Severity Diary (DGSSD), recorded in an electronic diary (e-diary). The DGSSS was derived as the sum of the weekly averages of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0=no or not at all uncomfortable to 10=worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period of the previous study or the run-in period of this study for new participants.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02 for rollover participants or Day -14 to Day -1 for new participants) to Week 12 of this study
Population: Modified-intent-to-treat (mITT) Population included all randomized participants with ≥1 postbaseline assessment of DGSSD. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 147 | 295
score on a scale
  Baseline | 20.3 (6.70) | 19.7 (6.39)
  Change from Baseline to Week 12: number analyzed (Participants) | 133 | 247
  Change from Baseline to Week 12 | -7.1 (8.82) | -6.5 (7.80)

2. Primary Outcome: Change From Baseline to Week 52 in the Weekly Average DGSSS
Description: Participants assessed the severity of diabetic gastroparesis symptoms daily using the DGSSD, recorded in an electronic diary (e-diary). The DGSSS was derived as the sum of the weekly averages of the 4 DGSSD items: nausea, abdominal pain, postprandial fullness and bloating. Each symptom was scored using an 11-point ordinal scale where: 0=no or not at all uncomfortable to 10=worst possible or most uncomfortable for a total possible DGSSS of 0 (best) to 40 (worst). The average weekly scores at Week 52 were the average of the DGSSS scores from Week 49 to Week 52. A negative change from Baseline indicates improvement. Baseline was defined as the average of the 2 weekly DGSSS from the run-in period of the previous study or the run-in period of this study for new participants.
Time Frame: Baseline (14-day Run-in Period of the previous relamorelin study RLM-MD-01 or RLM-MD-02 for rollover participants or Day -14 to Day -1 for new participants) to Week 52 of this study
Population: mITT Population included all randomized participants with ≥1 postbaseline assessment of DGSSD. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 147 | 295
score on a scale
  Baseline | 20.3 (6.70) | 19.7 (6.39)
  Change from Baseline to Week 52: number analyzed (Participants) | 65 | 129
  Change from Baseline to Week 52 | -10.7 (8.93) | -8.6 (8.92)

3. Primary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is an AE that begins or worsens after receiving study drug.
Time Frame: First dose of study drug to within 30 days of the last dose of study drug (Up to approximately 56 weeks)
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 145 | 299
Participants | 105 | 221

4. Primary Outcome: Number of Participants With Potential Clinically Significant (PCS) Clinical Laboratory Results
Description: Clinical Laboratory tests included Hematology, Chemistry and Urinalysis tests. The investigator determined if the results were clinically significant. Only those categories where at least 1 participant had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Up to 52 weeks
Population: Safety Population included all participants who received ≥1 administration of study treatment. Number analyzed is the number of participants with non-PCS Baseline values and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 145 | 299
Participants
  Hematocrit (RATIO): >1.1×Upper Limit of Normal Value (ULN): number analyzed (Participants) | 139 | 289
  Hematocrit (RATIO): >1.1×Upper Limit of Normal Value (ULN) | 0 | 1
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN): number analyzed (Participants) | 139 | 289
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN) | 5 | 14
  Hemoglobin (gram(g)/L): <0.9×LLN: number analyzed (Participants) | 137 | 288
  Hemoglobin (gram(g)/L): <0.9×LLN | 10 | 20
  Lymphocytes Absolute Cell Count (10^9/(Liter(L)): >1.5×ULN: number analyzed (Participants) | 141 | 287
  Lymphocytes Absolute Cell Count (10^9/(Liter(L)): >1.5×ULN | 1 | 5
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 141 | 287
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN | 2 | 9
  Mean Corpuscular Volume [femtoliter(fL)]: >1.1×ULN: number analyzed (Participants) | 140 | 284
  Mean Corpuscular Volume [femtoliter(fL)]: >1.1×ULN | 2 | 2
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 143 | 288
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN | 2 | 0
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 143 | 288
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN | 7 | 3
  Red Blood Cell Count (10^12/L):<0.9×LLN: number analyzed (Participants) | 141 | 290
  Red Blood Cell Count (10^12/L):<0.9×LLN | 2 | 10
  White Blood Cell Count (10^9/L): <0.7×LLN: number analyzed (Participants) | 144 | 291
  White Blood Cell Count (10^9/L): <0.7×LLN | 2 | 0
  Alanine Aminotransferase (Serum Glutamate-Pyruvate transaminase (SGPT)) (Unit (U)/L): ≥3.0×ULN: number analyzed (Participants) | 144 | 291
  Alanine Aminotransferase (Serum Glutamate-Pyruvate transaminase (SGPT)) (Unit (U)/L): ≥3.0×ULN | 0 | 6
  Albumin (gram (g)/L): <0.9×LLN: number analyzed (Participants) | 143 | 292
  Albumin (gram (g)/L): <0.9×LLN | 0 | 1
  Alkaline Phosphatase (U/L): ≥3.0×ULN: number analyzed (Participants) | 144 | 292
  Alkaline Phosphatase (U/L): ≥3.0×ULN | 0 | 1
  Aspartate Aminotransferase (Serum Glutamic-Oxaloacetic Transaminase (SGOT)) (U/L): ≥3.0×ULN: number analyzed (Participants) | 144 | 291
  Aspartate Aminotransferase (Serum Glutamic-Oxaloacetic Transaminase (SGOT)) (U/L): ≥3.0×ULN | 2 | 3
  Bicarbonate (HCO3) (millimole (mmol)/L): >1.1×ULN: number analyzed (Participants) | 138 | 290
  Bicarbonate (HCO3) (millimole (mmol)/L): >1.1×ULN | 3 | 2
  Bicarbonate (HCO3) (millimole (mmol)/L): >1.1×LLN: number analyzed (Participants) | 138 | 290
  Bicarbonate (HCO3) (millimole (mmol)/L): >1.1×LLN | 3 | 2
  Bicarbonate (HCO3) (millimole (mmol)/L): <0.9×LLN: number analyzed (Participants) | 138 | 290
  Bicarbonate (HCO3) (millimole (mmol)/L): <0.9×LLN | 6 | 6
  Bilirubin, Total (micromole (umol)/L): >1.5×ULN: number analyzed (Participants) | 144 | 292
  Bilirubin, Total (micromole (umol)/L): >1.5×ULN | 0 | 1
  Blood Urea Nitrogen (mmol/L): >1.2×ULN: number analyzed (Participants) | 125 | 272
  Blood Urea Nitrogen (mmol/L): >1.2×ULN | 14 | 27
  Calcium (mmol/L): >1.1×ULN: number analyzed (Participants) | 144 | 292
  Calcium (mmol/L): >1.1×ULN | 0 | 1
  Chloride (mmol/L): <0.9×LLN: number analyzed (Participants) | 144 | 292
  Chloride (mmol/L): <0.9×LLN | 1 | 1
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN: number analyzed (Participants) | 142 | 284
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN | 2 | 5
  Creatinine (umol/L): >1.3×ULN: number analyzed (Participants) | 134 | 275
  Creatinine (umol/L): >1.3×ULN | 15 | 20
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN: number analyzed (Participants) | 132 | 269
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN | 22 | 52
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN: number analyzed (Participants) | 132 | 269
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN | 4 | 14
  Glycohemoglobin A1C (%): Increase of ≥0.5%: number analyzed (Participants) | 144 | 292
  Glycohemoglobin A1C (%): Increase of ≥0.5% | 95 | 247
  Glycohemoglobin A1C (%): Increase of ≥1%: number analyzed (Participants) | 144 | 292
  Glycohemoglobin A1C (%): Increase of ≥1% | 94 | 246
  Phosphorus (mmol/L): >1.1×ULN: number analyzed (Participants) | 142 | 287
  Phosphorus (mmol/L): >1.1×ULN | 13 | 5
  Phosphorus (mmol/L): <0.9×LLN: number analyzed (Participants) | 142 | 287
  Phosphorus (mmol/L): <0.9×LLN | 1 | 4
  Potassium (mmol/L): <0.9×LLN: number analyzed (Participants) | 144 | 292
  Potassium (mmol/L): <0.9×LLN | 1 | 0
  Protein, Total (g)/L): >1.1×ULN: number analyzed (Participants) | 143 | 291
  Protein, Total (g)/L): >1.1×ULN | 1 | 0
  Triglycerides, Fasting (mmol/L): ≥3.0×ULN: number analyzed (Participants) | 140 | 280
  Triglycerides, Fasting (mmol/L): ≥3.0×ULN | 8 | 9
  Uric Acid (Urate) (umol/L): >1.1×ULN: number analyzed (Participants) | 114 | 233
  Uric Acid (Urate) (umol/L): >1.1×ULN | 17 | 37
  Uric Acid (Urate) (umol/L): <0.9×LLN: number analyzed (Participants) | 114 | 233
  Uric Acid (Urate) (umol/L): <0.9×LLN | 1 | 9

5. Primary Outcome: Number of Participants With Clinically Meaningful Trends for Vital Signs
Description: Vital Signs included assessments of heart rate, respiratory rate, systolic and diastolic blood pressure, and body temperature. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to 52 weeks
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 145 | 299
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Results
Description: A standard 12-lead ECG was performed. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to 52 weeks
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 145 | 299
Participants | 2 | 2

7. Primary Outcome: Number of Participants With a ≥1% Increase in Glycosylated Hemoglobin A1c (HbA1c)
Time Frame: Up to 52 weeks
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Relamorelin 10 μg
Number analyzed (Participants) | 145 | 299
Participants | 94 | 246

8. Primary Outcome: Number of Participants With Anti-relamorelin Antibody Testing Results by Visit
Description: A blood sample was collected that was sent to a laboratory for an anti-relamorelin antibody screening test. A positive screening test was confirmed by an immunodepletion assay. The number of participants in each of the following categories are reported: Negative Screening Test, Positive Screening Test, Negative Confirmatory Test, and Positive Confirmatory Test at each time point.
Time Frame: Baseline (Day 1), Day 84, Day 364, and End of Treatment (Up to Day 364)
Population: Safety Population included all participants who received ≥1 administration of double-blind study treatment (N=299 in the Relamorelin 10 μg arm). Anti-relamorelin antibody testing was only done for those participants who received treatment with relamorelin. Number analyzed is the number of participants with data available at the given timepoint. Due to a laboratory issue not all positive screening tests were confirmed.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin 10 μg
Number analyzed (Participants) | 299
Participants
  Screening Test (Baseline): number analyzed (Participants) | 166
  Screening Test (Baseline): Negative | 127
  Screening Test (Baseline): Positive | 39
  Confirmatory Test (Baseline): number analyzed (Participants) | 5
  Confirmatory Test (Baseline): Negative | 5
  Confirmatory Test (Baseline): Positive | 0
  Screening Test (Day 84): number analyzed (Participants) | 96
  Screening Test (Day 84): Negative | 73
  Screening Test (Day 84): Positive | 23
  Confirmatory Test (Day 84): number analyzed (Participants) | 7
  Confirmatory Test (Day 84): Negative | 6
  Confirmatory Test (Day 84): Positive | 1
  Screening Test (Day 364): number analyzed (Participants) | 14
  Screening Test (Day 364): Negative | 10
  Screening Test (Day 364): Positive | 4
  Confirmatory Test (Day 364): number analyzed (Participants) | 0
  Screening Test (End of Treatment): number analyzed (Participants) | 26
  Screening Test (End of Treatment): Negative | 20
  Screening Test (End of Treatment): Positive | 6
  Confirmatory Test (End of Treatment): number analyzed (Participants) | 1
  Confirmatory Test (End of Treatment): Negative | 1
  Confirmatory Test (End of Treatment): Positive | 0
  Screening Test (Unscheduled): number analyzed (Participants) | 3
  Screening Test (Unscheduled): Negative | 2
  Screening Test (Unscheduled): Positive | 1
  Confirmatory Test (Unscheduled): number analyzed (Participants) | 1
  Confirmatory Test (Unscheduled): Negative | 1
  Confirmatory Test (Unscheduled): Positive | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 30 days of the last dose of study drug (Up to approximately 56 weeks)
Description: All-Cause Mortality included all randomized participants. Adverse Events: Safety Population included all participants who received ≥1 administration of study treatment.
Arm/Group | Placebo | Relamorelin 10 μg
All-Cause Mortality (participants affected / at risk) | 0/148 | 2/302
Serious Adverse Events (participants affected / at risk) | 21/145 | 43/299
Other Adverse Events (participants affected / at risk) | 37/145 | 82/299
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Relamorelin 10 μg (N=299)
Cardiac arrest (Cardiac disorders) | 0 | 2
Acute left ventricular failure (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diabetic gastroparesis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Physical deconditioning (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 2 | 1
Bacteraemia (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Diabetic gangrene (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Relamorelin 10 μg (N=299)
Diarrhoea (Gastrointestinal disorders) | 14 | 21
Urinary tract infection (Infections and infestations) | 9 | 28
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 18
Headache (Nervous system disorders) | 7 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/46/NCT03383146/Prot_002.pdf
  • Statistical Analysis Plan (2020-12-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03383146/SAP_001.pdf